CLINICAL TRIAL: NCT03583866
Title: Adiposity and Endothelin Receptor Function
Acronym: END-RF
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ryan Harris, Assistant Professor, Augusta University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1148277; 5P01HL069999 (NIH)
Record Dates: First submitted 2018-06-27; First posted 2018-07-12 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: blood pressure; microdialysis
MeSH Terms: conditions — Hypertension | interventions — candesartan; candesartan cilexetil; Maltose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Candesartan (Experimental): Sub chronic (7 days) Candesartan (16 mg/day)
  Interventions: Drug: Candesartan
- Placebo (Placebo Comparator): Endothelial function will be determined following a seven day treatment of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Candesartan — 7 days of Candesartan (16mg/day)
  Other Names: Blopress, Atacand, Amias, and Ratacand
  Arms: Candesartan
Drug: Placebo — 7 days of Placebo
  Other Names: Lactose capsule, Maltose capsule
  Arms: Placebo

SUMMARY:
Elevated levels of ET-1 have been implicated in cardiovascular disease and some forms of hypertension. Due to the strong, positive correlation between obesity and hypertension, the present study will explore the contribution of adiposity in ETB receptor function and aim to elucidate if ETB receptor dysfunction is a major contributor to hypertension in obesity.

DETAILED DESCRIPTION:
The proposed study is designed to investigate the influence of adiposity on ETB receptor function and subsequent vascular responses. The combination of ET-1, ET-3, and the respective ETA and ETB receptor antagonists will be used to provide insight into the mechanisms of ETB receptor dysfunction in the presence of adiposity. Previous studies have revealed elevations in circulating ET-1 in obese individuals; therefore, we predict that obese subjects will exhibit 1) ETB receptor dysfuncton compared to lean subjects and 2) an improvement in ETB receptor dysfunction following treatment with Candesartan.

ELIGIBILITY:
Inclusion Criteria:

• If you are an adult between the ages of 18-40 year old

Exclusion Criteria:

* Evidence of cardiovascular, pulmonary, renal, hepatic, cerebral, or metabolic disease
* Evidence of pregnancy
* Using medications that affect vascular tone (i.e., nitrates, etc.)
* Use of any anticoagulants (i.e. aspirin)
* Anemia
* If you are postmenopausal
* If you have uncontrolled hypertension (treated resting SBP >140 mm Hg or DBP >90 mm Hg)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in Flow-Mediated Dilation (FMD) | pre-treatment Baseline and 7 days post-treatment
  Change in Brachial artery FMD induced by reactive hyperemia assessed vascular endothelial function at baseline and several hours after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Harris, PHD, CES, Principal Investigator — Augusta University
Locations (1):
- Georgia Prevention Institute/ Laboratory of Integrative and Exercise Physiology, Augusta, Georgia, United States

REFERENCES:
- See also: Laboratory of Integrative and Exercise Physiology Website — http://facebook.com/harrislab